CLINICAL TRIAL: NCT05310214
Title: Effect of Acupuncture and Laser Acupuncture on Pain and Functional Capacity in People With Chronic Nonspecific Low Back Pain: a Randomised Controlled, Blinded Clinical Trial
Brief Title: Effect of Acupuncture and Laser Acupuncture in the Treatment of People With Chronic Nonspecific Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fabiano Politti, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GA-2022
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Low Back Pain
Keywords: Acupuncture; laser therapy; low back pain; acupuncture points
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: randomised clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture treatment (ACP) (Experimental): The experimental group will be treated with acupuncture
  Interventions: Other: Acupuncture
- Laser acupuncture treatment (LACP) (Active Comparator): The active comparator group will be treated with laser acupuncture
  Interventions: Other: Laser acupuncture

INTERVENTIONS:
Other: Acupuncture — Treatment with ACP will be performed by inserting sterile acupuncture needles 0.25 x 13 mm into the acupoints BL23 (Shenshu), BL25 (Dachangshu), BL40 (Weizhong), BL62 (Qixue), SI3 (Houxi) and Jiaji , for the treatment of chronic non-specific low back pain. Interventions will last one hour, and will happen twice a week for 5 weeks.
  In order to increase the effectiveness of blinding for both groups, in this study the model was adopted: "combined simulated control". In this case, Sham acupuncture points will be used to simulate the treatment, as follows: i) Arms: 3 cm above the lateral epicondyle of the elbow, ii) Lumbar spine: Iliac crest on the same line as the greater trochanter of the femur. Thus, in the ACP group, the placebo LACP (without dosemetry) will be applied to these 4 points together with the real treatment.
  Arms: Acupuncture treatment (ACP)
Other: Laser acupuncture — The use of LACP (808 nm wavelength, 100 mW, energy 6 J per acp point), on acupoints BL23 (Shenshu), BL25 (Dachangshu), BL40 (Weizhong), BL62 (Qixue), SI3 (Houxi) and Jiaji will be used as a treatment for nonspecific chronic low back pain. Interventions will last one hour, and will happen twice a week for 5 weeks.
  Sham acupuncture points will be used to simulate the treatment, as follows: i) Arms: 3 cm above the lateral epicondyle of the elbow, ii) Lumbar spine: Iliac crest on the same line as the greater trochanter of the femur. These sham points will be inserted superficially so that the depth is sufficient to keep them fixed during the experiment, without individuals reporting the "dequi".
  Arms: Laser acupuncture treatment (LACP)

SUMMARY:
The aim of this randomized clinical trial will be to compare the efficacy between acupuncture and laser acupuncture on pain and disability in people with chronic nonspecific low back pain .

DETAILED DESCRIPTION:
Forty-four patients with chronic cnLBP of more than three months duration will be randomly allocated to two groups: acupuncture group (ACP) (n = 22) and laser acupuncture group (LACP) (n = 22).Interventions will last one hour, and will happen twice a week for 5 weeks. The primary clinical outcomes will be pain intensity (11-point numeric pain rating scale) as measured and functional disability (Oswestry Disability Index).The secondary outcomes will be the Pain Catastrophizing Scale, Patient-Specific Functional Scale and fingertip-to-floor test. Evaluations will be performed before and after the first session, after 5 weeks of treatment, and three months after randomization (follow-up). The findings will be analyzed statistically considering a 5% significance level (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Non-specific LBP for at least three months
* Pain intensity of at least 2 points measured using the Numeric Pain Rating Scale

Exclusion Criteria:

* Pregnancy;
* Any contraindication to ACP or having undergone treatment in the previous six months
* Having undergone spinal surgery in the previous six months;
* Serious spinal pathology (e.g. metastasis, spinal fracture, inflammatory, and infective diseases, caudal equine syndrome, canal stenosis, osteoporosis, rheumatoid arthritis and lumbar radiculopathy);
* Currently in an acute inflammatory phase of known gastrointestinal or urinary diseases (such as cholecysticis, renal calculi, peritonitis, appendicitis);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 3 months
  The Numeric Pain Rating Scale will be used to determine the level of pain intensity perceived by the patient using an 11-point scale on which 0 represents the absence of pain and 10 represents the worst pain imaginable.
Functional disability | 3 months
  The Oswestry Disability Index will be used to determine the functional disability of participants. Questionnaire examines perceived level of disability in 10 everyday activities of daily living. The 6 statements are scored from 0 to 5 with the first statement scoring 0 through to the last at 5. Interpretation of Scores
  1. 0% to 20% - minimal disability
  2. 21%-40% - moderate disability
  3. 41%-60%- severe disability
  4. 61%-80%- crippled
  5. 81%-100%: These patients are either bed-bound or exaggerating their symptoms.

SECONDARY OUTCOMES:
Pain Catastrophizing | 3 months
  The Pain Catastrophizing Scale will be used to assess catastrophic thinking related to pain. 13 items rated on 5-point Likert scales, from (0) not at all to (4) all the time. Higher score indicates higher level of catastrophizing
  Item scores are summed into a total score (PCS-T) and three subscale scores:
  * Rumination: Items 8, 9, 10, and 11 (response: 0-16 points)
  * Magnification: Items 6, 7, 13 (response: 0-12 points)
  * Helplessness: Items 1, 2, 3, 4, 5, and 12 (response: 0-24points) A total score above 30 indicates clinically relevant level of catastrophizing
Functional independence. | 3 months
  The Patient-Specific Functional Scale will be used to assess the participant's levels of functional independence. Patients are asked to rate (on an 11-point scale) the current level of difficulty associated with each activity. Following the intervention, patients are asked again to rate the activities previously identified (and are given the chance to nominate new problematic activities that might have arisen during that time).
  "0" represents "unable to perform" and "10" represents "able to perform at prior level"
Mobility of spine and pelvis | 3 months
  The fingertip-to-floor test will be used to evaluate the mobility of both the whole spine and the pelvis in the overall motion of bending forward.
  If the fingertip-to-floor test is "0"cm or the patient is able to place their palms to the floor with no pain, a different outcome measure should be considered.